CLINICAL TRIAL: NCT05746351
Title: Dexmedetomidine , Fentanyl or Nalbuphine As Additives to Epidural Bupivacaine for Labor Analgesia. A Double Blind Randomized Study.
Brief Title: Analgesic Additives to Epidural Bupivacaine in Normal Labor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abanob Fathy Zareef, Resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: epidural additives in labor
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Labor Pain
Keywords: epidural anathesia; normal labor
MeSH Terms: conditions — Labor Pain | interventions — Dexmedetomidine; Fentanyl; Nalbuphine

STUDY DESIGN:
Intervention Model Description: The participants will be divided into three equal groups ,one group will receive epidural analgesia with bupivacaine and dexmedetomidine, another Group will receive epidural analgesia with bupivacaine and fentanyl and the other Group will receive epidural analgesia with bupivacaine and Nalbuphine.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- epidural Bupivacaine with Dexmedetomidine in normal labor (Active Comparator): Epidural analgesia will be initiated and maintained using a solution of 0.125% bupivacaine with Dexmedetomidine 0.5 μg/ml
  Interventions: Drug: Dexmedetomidine
- epidural Bupivacaine with fentanyl in normal labor (Active Comparator): Epidural analgesia will be initiated and maintained using a solution of 0.125% bupivacaine with fentanyl 2 μg/ml.
  Interventions: Drug: fentanyl
- epidural Bupivacaine with Nalbuphine in normal labor (Active Comparator): Epidural analgesia will be initiated and maintained using a solution of 0.125% bupivacaine with 0.2 mg/ml Nalbuphine.
  Interventions: Drug: Nalbuphine

INTERVENTIONS:
Drug: Dexmedetomidine — a group will receive epidural Bupivacaine with Dexmedetomidine in normal labor
  Other Names: precedex
  Arms: epidural Bupivacaine with Dexmedetomidine in normal labor
Drug: fentanyl — a group will receive epidural Bupivacaine with fentanyl in normal labor
  Other Names: Durogesic
  Arms: epidural Bupivacaine with fentanyl in normal labor
Drug: Nalbuphine — a group will receive epidural Bupivacaine with Nalbuphine in normal labor
  Other Names: Nalufin
  Arms: epidural Bupivacaine with Nalbuphine in normal labor

SUMMARY:
The aim of the study will be to compare the role of Dexmedetomidine, Nalbuphine and fentanyl as additives to epidural bupivacaine in painless vaginal delivery as regard of effectiveness analgesia and maternal safety.

DETAILED DESCRIPTION:
Labor pain often causes a strong stress response. Several inhalation and parenteral anesthetics, sedatives, tranquilizers, and analgesics have been used for pain relief during labor, while over the last decade, lumbar epidural analgesia has greatly increased .

Recently, it was concerned by most mothers and doctors that how to alleviate the pain during delivery. The ideal labor analgesia should be based on maternal and child safety and should have a fast acting good analgesic effect and less adverse reaction .

Epidural anesthesia is convenient and has a less adverse reaction and obvious effect in the commonly used analgesic methods, which are widely used in the current way of analgesia .

Studies have confirmed the efficacy of dexmedetomidine in prolonging the duration of perineural nerve blocks. Specifically, perineural dexmedetomidine enhances sensory, motor, and analgesic block characteristics.

Dexmedetomidine is a selective α₂ receptor agonist and has a sympatholytic, sedative, and opioid sparing effect. It does not cause respiratory depression and can therefore be used as an adjuvant in certain clinical settings .

It has also been proved that dexmedetomidine would not increase the risk of side effects, such as nausea, headache, vomiting, shivering, and hypotension .

Nalbuphine is a synthetic agonist-antagonist opioid that has the characteristics of Mu-antagonist and Kappa-agonist activities. Nalbuphine has gained parenteral analgesia for intraoperative, postoperative, and obstetrical uses .

The analgesic potency of nalbuphine has been found to be equal to morphine, but unlike morphine, it shows a ceiling effect on respiratory depression. It has the potential to provide effective postoperative analgesia with no risk of respiratory depression .

ELIGIBILITY:
Inclusion Criteria:

* >/= 18 years of age
* American Society of Anesthesiologists (ASA) Physical Status 2 or 3
* Full term pregnancy (>37 gestational weeks)
* Planning vaginal delivery
* Planning epidural labor analgesia
* Vertex presentation

Exclusion Criteria:

* Patient refusal to epidural analgesia,
* Contraindications of epidural analgesia (coagulopathy, local infection, vertebral deformity)
* Allergy to study agents (hypersensitivity to bupivacaine, Nalbuphine, fentanyl or dexmedetomidine)
* hemodynamic instability, severe aortic or mitral stenosis)
* Severe pre-eclampsia,
* Breech presentations
* Antepartum hemorrhage
* Cephalopelvic disproportion
* Body mass index ≥40 kg/m2.
* Uncontrolled systemic comorbidities [i.e., diabetes, hepatic, renal or cardiac]
* Known or suspected fetal abnormalities
* Inability to communicate or participate in study procedures

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 69 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
VAS score for pain | before epidural analgesia, 30 minutes from time 0, at 1 hour and hourly till end of 3rd stage of delivery.
  changes in VAS score for pain before epidural analgesia, 30 minutes from time 0, at 1 hour and hourly till end of 3rd stage of delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Zein EA Zareh Hassan, professor, Study Chair — Assiut University; Elwani Eldramy Elsenosi, professor, Study Director — Assiut University; Khaled Tolba Younes, Lecturer, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Paramasivan A, Lopez-Olivo MA, Foong TW, et al. Intrathecal dexmedetomidine and postoperative pain: a systematic review and meta-analysis of randomized controlled trials. Eur J Pain. 2020;24(7):1215-1227 — https://pubmed.ncbi.nlm.nih.gov/32333825/
- See also: Senapati LK, Samanta P. Effect of intravenous versus intrathecal dexmedetomidine on characteristics of hyperbaric bupivacaine spinal anesthesia in lower limb surgery. Asian J Pharm Clin Res. 2018;11:427-430. — https://innovareacademics.in/journals/index.php/ajpcr/article/view/26096
- See also: Santpur MU, Kahalekar GM, Saraf N, et al. Effect of intravenous dexmedetomidine on spinal anesthesia with 0.5% hyperbaric bupivacaine in lower abdominal surgeries: a prospective randomized control study. Anesth Essays Res. 2016;10(3):497-501. — https://pubmed.ncbi.nlm.nih.gov/27746540/
- See also: ] Niu XY, Ding XB, Guo T, et al. Effects of intravenous and intrathecal dexmedetomidine in spinal anesthesia: a meta-analysis. CNS Neurosci Ther. 2013;19(11):897-904. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6493572/
- See also: Camann WR, Hurley RH, Gilbertson LI, et al. Epidural nalbuphine for analgesia following caesarean delivery: dose-response and effect of local anaesthetic choice. Can J Anaesth. 1991;38(6):728-732. — https://pubmed.ncbi.nlm.nih.gov/1914055/
- See also: ] Chatrath V, Attri JP, Bala A, et al. Epidural nalbuphine for postoperative analgesia in orthopedic surgery. Anesth Essays Res. 2015;9(3):326. — https://pubmed.ncbi.nlm.nih.gov/26712968/